CLINICAL TRIAL: NCT00484016
Title: Drug Delivery and Toxicities of Adjuvant Chemotherapy in Resected Non Small Cell Lung Cancer
Brief Title: Drug Delivery and Toxicities of Adjuvant Chemotherapy in Resected NCSLC
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0155
Record Dates: First submitted 2007-06-04; First posted 2007-06-08 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Adjuvant; Chemotherapy; Lung; Cancers
Keywords: adjuvant; chemotherapy; observation; resected; cancers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There are limited numbers of retrospective studies showing the effectiveness of adjuvant chemotherapy over observation in resected lung cancers.

DETAILED DESCRIPTION:
We propose to retrospectively examine the Washington University School of Medicine experience on all patients receiving adjuvant chemotherapy between 2003 and 2005. We will retrospectively analyze the survival and outcomes in the lung cancer patients receiving adjuvant chemotherapy following surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received adjuvant chemotherapy
* 18-88 years

Exclusion Criteria:

* Any patients that have not received adjuvant chemotherapy
* Patients under 18 or over 88

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Result] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu